CLINICAL TRIAL: NCT01885299
Title: Multi-Institution Registry of SRS/SBRT Procedures
Brief Title: RSSearch Patient Registry-Long Term Study of Use of SRS/SBRT
Status: Recruiting | Type: Observational
Sponsor: The Radiosurgery Society (Other)
Collaborators: VisionTree (Unknown)
Responsible Party: Sponsor
Other Study IDs: RSSearch Patient Registry; NCT01563549 (obsolete NCT alias)
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Neoplasms; Arteriovenous Malformation of Central Nervous System; Trigeminal Neuralgia
Keywords: Radiosurgery; CyberKnife; Benign tumors; Malignant tumors; Cranial tumors; Extracranial tumors; Lung; Liver; Pancreas; Prostate; Stereotactic radiosurgery; Stereotactic body radiotherapy
MeSH Terms: conditions — Neoplasms; Trigeminal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients being treated by SRS/SBRT: Patients with a condition being considered for treatment by SRS/SBRT
  Interventions: Radiation: SRS/SBRT

INTERVENTIONS:
Radiation: SRS/SBRT — Intervention varies by condition being treated.

SUMMARY:
The RSSearch® Registry is an international multi-year database designed to track SRS/SBRT (Stereotactic Radiosurgery/Stereotactic Body Radiation Therapy) utilization, treatment practices and outcomes to help determine, over time, the most effective use of these systems in management of patients with life threatening tumors and other diseases. (This study was formally called ReCKord and included the CyberKnife only; The ReCKord study continues as a CyberKnife subset of RSSearch.)

DETAILED DESCRIPTION:
The Registry is designed to help SRS/SBRT (Stereotactic Radiosurgery/Stereotactic Body Radiation Therapy) users to understand utilization of and key treatment outcomes for these treatment approaches. Some of the objectives include:

Allow participants to record information about usage of SRS/SBRT in everyday practice, including patient characteristics and disease information, treatment plans and outcomes Provide participants with ready access to data for publication of their own experience and as a tool for establishing collaborations with other participating sites Facilitate quality improvement efforts for individual treatment providers Understand the effectiveness of different treatment plans for different types of lesions, diseases and treatments

The Registry tracks select outcomes for each condition treated by SRS/SBRT (for example, PSA for prostate cancer); the Registry also provides individual participants the ability to add additional outcomes for each and any condition of specific interest to their institutions.

The Registry is hosted by Vision Tree, Inc who is an independent vendor of electronic registries; they are responsible for HIPAA compliance, including all security mechanisms.

Patients will be enrolled prospectively. Some retrospective patient data is likely to be included in order to capture both short and longer term outcomes data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of benign or malignant tumors or other conditions deemed treatable by stereotactic radiosurgery or stereotactic body radiotherapy
* Willingness to sign an Informed Consent Document or verbally agree to participation

Exclusion Criteria:

* There are no specific exclusion criteria, but patients who are unwilling to sign the ICD or who decline participation will not be included

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patients who have a SRS/SBRT procedure
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2012-03; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years
  Survival from time of treatment to death

SECONDARY OUTCOMES:
Local and distant recurrence | One to Five years
  Calculated from time of treatment to recurrence

OTHER OUTCOMES:
Treatment toxicity | Immediate -5 years
  Complications of treatment. These complications are organ specific depending on which organ is being treated. For example, if the prostate is being treated,there may be rectal and urinary complications. If the brain is being treated, there may be headaches or nausea. The Radiation Therapy Oncology Group (RTOG) scale used for defining and measuring complications of radiotherapy is incorporated into the Registry database.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Mahadevan, MD, Study Director — The Radiosurgery Society
Locations (13):
- United States (13):
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Sylvester Comprehensive Cancer Center, University of Miami, Miami, Florida
  - Southeast Georgia Health System, Brunswick, Georgia
  - Henry Ford Health System, Detroit, Michigan
  - AtlantiCare Regional Medical Center and AtlantiCare Cancer Care Institute, Egg Harbor, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - NJ Cyberknife at Community Medical Center, Toms River, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Geisinger Health System, Danville, Pennsylvania
  - Philadelphia CyberKnife, Philadelphia, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Cyberknife at Erlanger, Chattanooga, Tennessee
  - St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Background] Tipton KN, Sullivan N, Bruening W, Inamdar R, Launders J, Uhl S, Schoelles KM. Stereotactic Body Radiation Therapy [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2011 May. Report No.: 10(11)-EHC058-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK55723/ PMID 21735562
- [Background] Dieterich S, Gibbs IC. The CyberKnife in clinical use: current roles, future expectations. Front Radiat Ther Oncol. 2011;43:181-194. doi: 10.1159/000322423. Epub 2011 May 20. PMID 21625154
- [Background] Wowra B, Muacevic A, Tonn JC. CyberKnife radiosurgery for brain metastases. Prog Neurol Surg. 2012;25:201-9. doi: 10.1159/000331193. Epub 2012 Jan 6. PMID 22236681
- [Background] Sarwate D, Sarkar S, Krimsky WS, Burgan CM, Patel K, Evans R, Harley DP. Optimization of mediastinal staging in potential candidates for stereotactic radiosurgery of the chest. J Thorac Cardiovasc Surg. 2012 Jul;144(1):81-6. doi: 10.1016/j.jtcvs.2012.03.004. Epub 2012 Apr 11. PMID 22498085
- [Background] Sohn S, Chung CK. The role of stereotactic radiosurgery in metastasis to the spine. J Korean Neurosurg Soc. 2012 Jan;51(1):1-7. doi: 10.3340/jkns.2012.51.1.1. Epub 2012 Jan 31. PMID 22396835
- [Background] Davis JN, Medbery C, Sharma S, Pablo J, Kimsey F, Perry D, Muacevic A, Mahadevan A. Stereotactic body radiotherapy for centrally located early-stage non-small cell lung cancer or lung metastases from the RSSearch((R)) patient registry. Radiat Oncol. 2015 May 15;10:113. doi: 10.1186/s13014-015-0417-5. PMID 25975848
- [Background] Davis JN, Medbery C 3rd, Sharma S, Perry D, Pablo J, D'Ambrosio DJ, McKellar H, Kimsey FC, Chomiak PN, Mahadevan A. Stereotactic body radiotherapy for early-stage non-small cell lung cancer: clinical outcomes from a National Patient Registry. J Radiat Oncol. 2015;4(1):55-63. doi: 10.1007/s13566-014-0177-0. Epub 2015 Jan 31. PMID 25774243
- [Background] Davis JN, Medbery C 3rd, Sharma S, Danish A, Mahadevan A. The RSSearch Registry: patterns of care and outcomes research on patients treated with stereotactic radiosurgery and stereotactic body radiotherapy. Radiat Oncol. 2013 Nov 25;8:275. doi: 10.1186/1748-717X-8-275. PMID 24274599
- [Background] Ricco A, Davis J, Rate W, Yang J, Perry D, Pablo J, D'Ambrosio D, Sharma S, Sundararaman S, Kolker J, Creach KM, Lanciano R. Lung metastases treated with stereotactic body radiotherapy: the RSSearch(R) patient Registry's experience. Radiat Oncol. 2017 Feb 1;12(1):35. doi: 10.1186/s13014-017-0773-4. PMID 28143558
- [Background] Davis J, Sharma S, Shumway R, Perry D, Bydder S, Simpson CK, D'Ambrosio D. Stereotactic Body Radiotherapy for Clinically Localized Prostate Cancer: Toxicity and Biochemical Disease-Free Outcomes from a Multi-Institutional Patient Registry. Cureus. 2015 Dec 4;7(12):e395. doi: 10.7759/cureus.395. PMID 26798571
- [Background] Singh R, Davis J, Sharma S. Stereotactic Radiosurgery for Trigeminal Neuralgia: A Retrospective Multi-Institutional Examination of Treatment Outcomes. Cureus. 2016 Apr 3;8(4):e554. doi: 10.7759/cureus.554. PMID 27182468
- [Derived] Mahadevan A, Blanck O, Lanciano R, Peddada A, Sundararaman S, D'Ambrosio D, Sharma S, Perry D, Kolker J, Davis J. Stereotactic Body Radiotherapy (SBRT) for liver metastasis - clinical outcomes from the international multi-institutional RSSearch(R) Patient Registry. Radiat Oncol. 2018 Feb 13;13(1):26. doi: 10.1186/s13014-018-0969-2. PMID 29439707

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT01885299/Prot_ICF_000.pdf